CLINICAL TRIAL: NCT06321263
Title: Comparison of the Effects of Peripheral Muscle Training and Inspiratory Muscle: Randomized Clinical Study.
Brief Title: Comparison of the Effects of Peripheral Muscle Training and Inspiratory Muscle Training in Geriatric Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Associate professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 798307
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Muscle Strength
Keywords: Muscle strength; Physical performance; Respiratory muscle strength; Functional capacity; Quality of life

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peripheral Muscle Training Group (Experimental): Older individuals in this group will participate in group exercise training, including aerobic and resistance training, twice a week for ten weeks, each session supervised by a researcher physiotherapist and lasting one hour.
  Interventions: Other: Peripheral Muscle Training and step aerobics training
- Inspiratory Muscle Training Group: (Experimental): Older people in this group will perform aerobic and resistance training for 1 hour a day, twice a week for ten weeks, under the supervision of a researcher physiotherapist. As for Inspiratory Muscle Training, they will participate in training with 30 breathing cycles a day, six days a week, for ten weeks (two days in the clinic, four days at home).
  Interventions: Other: Inspiratory Muscle Training and step aerobics training

INTERVENTIONS:
Other: Peripheral Muscle Training and step aerobics training — First 5-minute warm-up in the protocol (calisthenic exercises); 30-40 minutes of resistance exercises and step aerobic exercises and the last 5 minutes cooling (stretching exercises) period will be applied.
  Other Names: Peripheral Muscle Training
  Arms: Peripheral Muscle Training Group
Other: Inspiratory Muscle Training and step aerobics training — First 5-minute warm-up in the protocol (calisthenic exercises); 30-40 minutes of resistance exercises and step aerobic exercises and the last 5 minutes cooling (stretching exercises) period will be applied.
  Other Names: Inspiratory Muscle Training
  Arms: Inspiratory Muscle Training Group:

SUMMARY:
In geriatric individuals, there is a decrease in muscle strength, muscle mass and physical performance with ageing. These physiological changes occurring in geriatric individuals make maintaining the physical activity necessary for a healthy life difficult. Weakness of respiratory muscles in geriatric individuals can increase the prevalence of diseases and disability. It has been shown in the literature that peripheral muscle training and inspiratory muscle training increase exercise capacity similarly. The effectiveness of moderate-intensity peripheral muscle training and inspiratory muscle training in sarcopenic geriatric individuals was compared and found to have similar effects on muscle strength.

Our study aims to compare the effects of inspiratory and peripheral muscle training in addition to aerobic exercise on muscle strength, physical performance, respiratory muscle strength, functional capacity, sarcopenia, and quality of life.

DETAILED DESCRIPTION:
Aging causes decline in physiological systems, including the cardiorespiratory system, musculo-skeletal system, vestibulo-ocular system, slowed postural control and cognitive function (especially dual task and executive functions). These changes occurring in geriatric individuals are an increased risk factor for various diseases and affect the individual's daily living activities, working life, addiction status and communication with the environment.

The most recommended physical activity subgroups in the guidelines for geriatric individuals are aerobic exercises, strengthening exercises, flexibility exercises and balance exercises. Physiological changes that occur in the organism during the aging process can cause muscle weakness, functional losses/limitations, balance problems, cognitive problems, chronic diseases and mortality. However, physiological and mechanical respiratory changes in geriatric individuals; It is known that there is a decrease in lung elasticity, respiratory muscle strength and chest wall compliance. These physiological changes make it difficult to maintain the physical activity necessary for a healthy life. It has also been shown that weakness of respiratory muscles in geriatric individuals can increase the rate of morbidity and mortality.

It is reported in the literature that respiratory muscle training (RMT) strengthens the diaphragm in geriatric individuals and may have a protective effect against respiratory tract infections by improving aerobic capacity, physical performance and coughing skill. In addition, studies have shown that Inspiratory Muscle Training (IMT) increases the strength of the inspiratory respiratory muscles, allows a more mechanically effective breathing pattern, and provides improvements in exercise capacity, diaphragm thickness and mobility, cardiac autonomic control and functional autonomy. Studies have shown that IMT is effective and applicable in improving balance ability. It has been reported to improve dynamic and reactive balance, as well as gait speed and inspiratory muscle function in healthy geriatric individuals. Considering the stated benefits of IMT, some authors suggest that it is an alternative or complementary training method that can be used for geriatric individuals, especially when other types of exercise are not possible, and that it should be added to rehabilitation programs.

In general, it has been reported in the literature that resistant exercise training is preferred as an intervention in geriatric individuals and that this training improves muscle strength, physical performance and functional performance. In a study where a high-intensity resistance training program was applied in sarcopenic geriatric women, it was reported that it increased respiratory muscle strength and Maximum Expiratory Pressure (MEP) and affected health-related quality of life.

There are opinions reported in the literature that improvement in peripheral and inspiratory muscle strength will reduce the risk of mortality. The effects of moderate-intensity peripheral muscle training and inspiratory muscle training were compared in sarcopenic geriatric individuals and were found to have similar effects on muscle strength. It has been reported that there is no significant change in muscle mass and physical performance. However, no study has been found in which the aerobic and strengthening exercises recommended for geriatric individuals are combined. In order to shed light on this deficiency in the literature, the investigators aim in our study to compare the effects of peripheral muscle training and inspiratory muscle training combined with aerobic training on muscle strength, physical performance, functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 65 years to 80 years (Older ),
* Standardised Mini Mental Test score ≥ 20,
* To walk 10 meters with or without an assistive device,
* If the participants answered No all of the questions of The Physical Activity Readiness Questionnaire
* Volunteering to participate in the study

Exclusion Criteria:

* With serious neurological and orthopedic problems that may prevent them from exercising,
* With serious vision and hearing problems,
* With a psychiatric disease,
* With serious cardiac and pulmonary system diseases that may prevent them from exercising,
* With vestibular system problems or medication use that may affect the vestibular system,
* Smokers.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The sociodemographic data form | Ten weeks
  Socio-demographic data of individuals (name-surname, age, gender, height,weight, smoking, occupation, education) will be collected with the demographic data collection form created by the researchers. In the clinical information section, other diseases and medications used will be recorded.
Hand grip strength | Ten weeks
  Three consecutive measurements will be made on the dominant hand with a Jamar hand dynamometer, 1 minute apart, and the highest value will be recorded.
Maximal inspiratory and expiratory pressures (MIP, MEP) | Ten weeks
  Static inspiratory (MIP) or expiratory (MEP) mouth pressures assess respiratory muscle strength.
6-Minute Walk Test (6MWT) | Ten weeks
  The 6MWT will be used to measure functional capacity.
The Short Physical Performance Battery (SPPB) | Ten weeks
  SPPB is a set of tests that combine gait speed, chair stand, and balance measures. It is used to predict possible disability and monitor function in older individuals.
Assessment of seniors᾽ quality of life: WHOQOL-OLD questionnaire | Ten weeks
  WHOQOL-OLD, a 24-item QOL measure, was developed by the WHOQOL Group as an add-on module to their QOL measures, specifically for use with older adults. A total score is the mean of the summed facet scores and ranges from one to five, with higher scores indicating better QOL.

SECONDARY OUTCOMES:
SARC-F questionnaire | Ten weeks
  It is a rapid diagnostic test developed for sarcopenia. A SARC-F survey score ≥ 4 is important for the diagnosis of sarcopenia. SARC-F score range is from 0 to 10; 0-3 points represent healthy condition, 4 points and above represent symptomatic condition.

OTHER OUTCOMES:
Canadian Occupational Performance Measure | Ten weeks
  The COPM will be used to identify the individual's activity performance problems and measure performance and satisfaction levels. A difference of 2 points from pre-test to post-test on either performance or satisfaction represents a clinically significant difference on the COPM.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akıncı, Ass.Prof., Study Director — Biruni University; Sezen Uyanık, MSc, Principal Investigator — Çanakkale Onsekiz Mart University
Locations (1):
- Golden Years Life Center, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Ferraro FV, Gavin JP, Wainwright TW, McConnell AK. Comparison of balance changes after inspiratory muscle or Otago exercise training. PLoS One. 2020 Jan 24;15(1):e0227379. doi: 10.1371/journal.pone.0227379. eCollection 2020. PMID 31978126
- [Background] Flor-Rufino C, Barrachina-Igual J, Perez-Ros P, Pablos-Monzo A, Martinez-Arnau FM. Resistance training of peripheral muscles benefits respiratory parameters in older women with sarcopenia: Randomized controlled trial. Arch Gerontol Geriatr. 2023 Jan;104:104799. doi: 10.1016/j.archger.2022.104799. Epub 2022 Aug 29. PMID 36070636
- [Background] Hallage T, Krause MP, Haile L, Miculis CP, Nagle EF, Reis RS, Da Silva SG. The effects of 12 weeks of step aerobics training on functional fitness of elderly women. J Strength Cond Res. 2010 Aug;24(8):2261-6. doi: 10.1519/JSC.0b013e3181ddacc6. PMID 20634751
- [Background] Cebria I Iranzo MA, Balasch-Bernat M, Tortosa-Chulia MA, Balasch-Parisi S. Effects of Resistance Training of Peripheral Muscles Versus Respiratory Muscles in Older Adults With Sarcopenia Who are Institutionalized: A Randomized Controlled Trial. J Aging Phys Act. 2018 Oct 1;26(4):637-646. doi: 10.1123/japa.2017-0268. Epub 2018 Aug 27. PMID 29431561
- [Background] Joung HJ, Lee Y. Effect of Creative Dance on Fitness, Functional Balance, and Mobility Control in the Elderly. Gerontology. 2019;65(5):537-546. doi: 10.1159/000499402. Epub 2019 May 3. PMID 31055579
- [Background] Kalapotharakos VI, Diamantopoulos K, Tokmakidis SP. Effects of resistance training and detraining on muscle strength and functional performance of older adults aged 80 to 88 years. Aging Clin Exp Res. 2010 Apr;22(2):134-40. doi: 10.1007/BF03324786. PMID 20440099
- [Background] Kim SH, Shin MJ, Lee JM, Huh S, Shin YB. Effects of a new respiratory muscle training device in community-dwelling elderly men: an open-label, randomized, non-inferiority trial. BMC Geriatr. 2022 Feb 24;22(1):155. doi: 10.1186/s12877-022-02828-8. PMID 35209851
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Background] Power M, Quinn K, Schmidt S; WHOQOL-OLD Group. Development of the WHOQOL-old module. Qual Life Res. 2005 Dec;14(10):2197-214. doi: 10.1007/s11136-005-7380-9. PMID 16328900
- [Background] Puthoff ML. Outcome measures in cardiopulmonary physical therapy: short physical performance battery. Cardiopulm Phys Ther J. 2008 Mar;19(1):17-22. No abstract available. PMID 20467494
- [Background] Segev-Jacubovski O, Herman T, Yogev-Seligmann G, Mirelman A, Giladi N, Hausdorff JM. The interplay between gait, falls and cognition: can cognitive therapy reduce fall risk? Expert Rev Neurother. 2011 Jul;11(7):1057-75. doi: 10.1586/ern.11.69. PMID 21721921
- [Background] Seixas MB, Almeida LB, Trevizan PF, Martinez DG, Laterza MC, Vanderlei LCM, Silva LP. Effects of Inspiratory Muscle Training in Older Adults. Respir Care. 2020 Apr;65(4):535-544. doi: 10.4187/respcare.06945. Epub 2019 Oct 29. PMID 31662444
- [Background] Woo J, Leung J, Morley JE. Validating the SARC-F: a suitable community screening tool for sarcopenia? J Am Med Dir Assoc. 2014 Sep;15(9):630-4. doi: 10.1016/j.jamda.2014.04.021. Epub 2014 Jun 16. PMID 24947762